CLINICAL TRIAL: NCT03743675
Title: Influence of Aerobic Training and Weight Loss on Skeletal Muscle Inflammatory Markers
Brief Title: Influence of Aerobic Training and Weight Loss on Skeletal Muscle Inflammatory Markers and Muscle Protein Balance in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miami University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: #01488r
Record Dates: First submitted 2018-10-18; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Overweight and Obesity; Inflammation; Muscle; Sedentary Lifestyle
Keywords: Overweight; Exercise Training; Older Adults; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Myositis, Inclusion Body; Sedentary Behavior; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diet-Induced Weight Loss (Experimental): Subjects in this arm will undergo 6-months of dietary counseling targeting 5-10% weight loss by the end of the intervention period.
  Interventions: Behavioral: Diet-Induced Weight Loss
- Exercise Training (Experimental): Subjects in this arm will undergo 6-months of supervised aerobic exercise training (3 days per week, moderate-to-vigorous intensity).
  Interventions: Behavioral: Aerobic Exercise Training
- Diet Plus Exercise (Experimental): Subjects in this arm will undergo 6-months of dietary counseling targeting 5-10% weight loss by the end of the intervention period. They will simultaneously undergo 6-months of supervised aerobic exercise training (3 days per week, moderate-to-vigorous intensity).
  Interventions: Behavioral: Diet-Induced Weight Loss; Behavioral: Aerobic Exercise Training
- Control (No Intervention): Subjects in this group will be asked to maintain their habitual physical activity, and will received counseling regarding a healthy, weight-maintenance diet.

INTERVENTIONS:
Behavioral: Diet-Induced Weight Loss — Diet-Induced Weight Loss: The goal of the diet intervention is to produce a weight loss of approximately 5-10% of body weight over the six-month period, which is consistent with the goals for obesity treatment outlined by the Academy of Nutrition and Dietetics (AND). According to the 2016 AND position paper for obesity-related interventions, this level of weight loss produces clinically significant reductions in biometrics (biochemical and anthropometrics measurements) and associated risk factors for chronic disease. Additionally, obese older adults who achieve weight loss intentionally through lifestyle changes experience improved physical function. This intervention will last for 6-months with bi-weekly face-to-face counseling sessions with a registered dietitian.
  Arms: Diet Plus Exercise; Diet-Induced Weight Loss
Behavioral: Aerobic Exercise Training — Exercise Intervention: Subjects will exercise on a cycle ergometer during the training sessions. Each session will consist of 1) a 5-10 minute warm up at "light" intensity; 2) a 20 to 30-minute training phase at "moderate-to-vigorous" intensity; and 3) a 5-minute cool down phase at "light". The training will be conducted 3 days per week for 6 months.
  Arms: Diet Plus Exercise; Exercise Training

SUMMARY:
It is estimated that 15% of adults aged 60-70 years, and up to 50% of adults aged 80 years and older are affected by sarcopenia-the age related loss of muscle mass and function. A disruption of the homeostatic balance between periods of muscle protein breakdown (predominant during fasting) and muscle protein synthesis (predominant following nutrient ingestion) can result in the loss of muscle mass over time. In particular, research suggests that an inability of muscle to fully respond to the anabolic influence of nutrient intake may contribute significantly to age-related muscle loss. This anabolic resistance is likely influenced by increased age-related inflammation. There is evidence in cell line and animal models that increased levels of the inflammatory cytokine, tumor necrosis factor-α (TNFα) impairs the molecular pathways that initiate muscle protein synthesis (i.e. mammalian target of rapamycin, mTOR signaling), and can accelerate muscle protein breakdown. Obesity, and sedentary lifestyle have been linked to increased TNFα expression, and thus may partially explain impaired muscle protein balance in older adults. The objectives of this clinical trial are to 1) determine if lifestyle modification via weight loss and aerobic exercise can reduce skeletal muscle inflammation and subsequently improve nutrient-stimulated muscle protein synthesis in previously sedentary, obese older adults; and 2) expose undergraduate Kinesiology and Nutrition majors to meritorious research. The investigators have recently published data with undergraduate researchers showing that body composition is associated with elevated skeletal muscle expression of TNFα converting enzyme (TACE). One of the primary actions of TACE is to cleave membrane bound TNFα (mTNFα) to soluble TNFα (sTNFα)-a more mature and bioactive form of TNFα. Both TACE and sTNFα are known to be elevated in a number of clinical conditions, including heart disease, cancer, arthritis, and diabetes. Based on these data, the investigators feel that TACE may represent an important and potentially modifiable (via weight loss and aerobic conditioning) regulator of skeletal muscle inflammation in humans. There are currently no data on the associations among skeletal muscle expression of TACE, TNFα, and muscle protein balance. Thus, the focus of this study is to determine if 5-10% diet-induced weight loss and 6-months (3 days per week) of aerobic exercise training can influence: 1) TACE and TNFα expression in skeletal muscle; and 2) improve molecular indices of muscle protein breakdown and nutrient-stimulated muscle protein synthesis (mTOR signaling) in sedentary, obese older adults. Specifically, 60 sedentary, obese older adults will be randomized to one of the following groups: 1) control group (CON), 2) a diet-induced weight loss group (DIET), 3) an aerobic exercise training group (EX), or 4) a diet-induced weight loss + aerobic exercise training group (DIET + EX). The results of this study will advance the understanding of the connections among skeletal muscle inflammation and muscle protein balance in older adults, and validate TACE as a potentially modifiable target for the prevention and treatment of sarcopenia and other age-related inflammatory diseases, which will contribute to the development of practice-based guidelines for healthcare practitioners.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 58 years or older
* Sedentary (<500 kcal/wk of physical activity)
* BMI > 30 kg/m2
* Stable body weight for at least 1 year
* Approval from primary care provider

Exclusion Criteria:

* Physical dependence
* History of falls (≥ 2/yr)
* Significant cardiovascular, metabolic, or pulmonary disease
* Implantable defibrillator or pacemaker
* Active cancer
* Recent (within 6 months) treatment with anabolic steroids, or corticosteroids
* Alcohol or drug abuse
* Prescription anti-coagulant use
* Allergy to lidocaine

Min Age: 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Inflammation | Change from baseline TACE and TNFa expression at 6 months
  Skeletal muscle biopsies will be taken at baseline and following 6-months of the interventions to assess changes in indices of inflammation including tumor necrosis factor-alpha (TNFa) and TNFa converting enzyme (TACE). Analyses will be made utilizing Western blots, along with appropriate loading and positive controls. Outcome data will be normalized to an internal loading control and presented as arbitrary units.
The activation of mammalian target of rapamycin (mTOR) signaling in the fasted and postprandial state | Change from baseline nutrient-stimulated mTOR and S6K1 activation at 6 months
  At baseline and following 6-months of the interventions, muscle biopsies will be taken in the fasted state and following ingestion of a beverage containing 0.5 g/kg body mass carbohydrate + 0.3 g/kg body mass protein by the subjects. 60 and 120 minutes after ingestion, biopsies will also be taken. Using Western blot analyses, the total and phosphorylated protein expression of mTOR, as well as its downstream signaling protein, S6K1 will be measured. Data will be expressed as phosphorylated-to-total abundance. This pathway has been shown to be critical for the stimulation of muscle protein synthesis (MPS) in response to nutrient intake. A higher ratio of phosphorylated:total abundance of these proteins (expressed as arbitrary units) indicates increased activation of MPS. It is hypothesized that the fasted-to-postprandial fold-change in activation of these proteins will be greater following 6-months of diet-induced weight loss and/or exercise training compared to a control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Miami University, Department of Kinesiology and Health, Phillips Hall, Oxford, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The investigators have no plans to make individual participant data available to researchers outside of their team.